CLINICAL TRIAL: NCT03720977
Title: Diagnostic Value and Biological Significant of cd71 in Lymphoid Dis Order
Brief Title: Diagnostic Value and Biological Significant of cd71 in Lymphoid Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marwa Aboelim Shafeik (Other)
Responsible Party: Sponsor-Investigator, Marwa Aboelim Shafeik, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: diagnostic value of cd71
Record Dates: First submitted 2018-10-18; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Lyphoid Disorders; cd71

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CD71 is expressed on activated B and T cells, macrophages, reticulocytes, erythroid precursors, and malignant tissues. , reflecting the requirement for iron in hemoglobin. , CD71 expression is upregulated on immature proliferating cells and low levels on resting mature lymphocytes. In addition to this general function, CD71 appears to play a costimulatory role in T cell activation and receptor for IgA1 antibodies So it is growth receptor that may help in diagnosis of lymphoid disorder and in differentiation of malignant and benign that will be studied investigate CD71 expression in lymphoid disorders and its diagnostic value ,we from collect data patient and do rotune examination

DETAILED DESCRIPTION:
1. Routine investigations for diagnosis:

   * CBC.
   * Bone marrow aspiration morphology.
   * Cytochemistry.
   * Flow cytometry immunophenotyping.
   * Bone marrow biopsy when indicated.
2. Special investigation is flow cytometry examination of CD71 expression.

sample size calculation ; sample size cases 39 sample size controls 39 total sample size 79 sample will be collected from patient in hospital university ,Data will be analysed by SPSS program

ELIGIBILITY:
Inclusion Criteria:

* all patients wiil be diagnosed lymphoid disorders

Exclusion Criteria:

* not present

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: confidence level 95 sample size 139
Sampling Method: Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
determin diagnostic value of cd71 in lymphoid disorder | baseline
  Routine investigations for diagnosis:
  CBC. Bone marrow aspiration morphology. Cytochemistry. Flow cytometry immunophenotyping. Bone marrow biopsy when indicated. Special investigation is flow cytometry examination of CD71 expression.
  total sample size 79 person .sample will be collected from patient in hospital university ,Data will be analysed by SPSS program it is growth receptor is expressed on activated B and T cells, macrophages, reticulocytes, erythroid precursors, and malignant tissues

CONTACTS AND LOCATIONS:
Overall Officials: Maged Salah, Prof, Study Director — Assiut University .clinical pathologydepartment

IPD SHARING:
Plan to Share IPD: No
immunophenotyping by flow cytometry of cd71

REFERENCES:
- [Background] Zhang Q, Steensma DP, Yang J, Dong T, Wu MX. Uncoupling of CD71 shedding with mitochondrial clearance in reticulocytes in a subset of myelodysplastic syndromes. Leukemia. 2019 Jan;33(1):217-229. doi: 10.1038/s41375-018-0204-z. Epub 2018 Jul 26. PMID 30050123
- [Background] Salzberger W, Martrus G, Bachmann K, Goebels H, Hess L, Koch M, Langeneckert A, Lunemann S, Oldhafer KJ, Pfeifer C, Poch T, Richert L, Schramm C, Wahib R, Bunders MJ, Altfeld M. Tissue-resident NK cells differ in their expression profile of the nutrient transporters Glut1, CD98 and CD71. PLoS One. 2018 Jul 20;13(7):e0201170. doi: 10.1371/journal.pone.0201170. eCollection 2018. PMID 30028872
- [Result] Dunsmore G, Koleva P, Ghobakhloo N, Sutton R, Ambrosio L, Meng X, Hotte N, Nguyen V, Madsen KL, Dieleman LA, Huang V, Elahi S. Lower Abundance and Impaired Function of CD71+ Erythroid Cells in Inflammatory Bowel Disease Patients During Pregnancy. J Crohns Colitis. 2019 Feb 1;13(2):230-244. doi: 10.1093/ecco-jcc/jjy147. PMID 30272151